CLINICAL TRIAL: NCT04369027
Title: Can Dynamic Changes of Pulse Pressure Variation During Passive Leg Raising or a Tidal Volume Challenge Help Predicting Preload Responsiveness in Mechanically Ventilated Patients With Spontaneous Breathing Activity
Brief Title: Changes of Pulse Pressure Variation Duing Tidal Volume Challenge in Patients With Spontaneous Breathing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Antoine Beclere (Other)
Responsible Party: Principal Investigator, Hamzaoui Olfa, PRINCIPAL INVESTIGATOR, Hopital Antoine Beclere
Other Study IDs: 2018-A00727-48
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preload responders: patients who increase their delta VTI by more than 10% during PLR
  Interventions: Diagnostic Test: passive leg raising
- preload unresponders: patients who do not increase their delta VTI by more than 10% during PLR

INTERVENTIONS:
Diagnostic Test: passive leg raising — passive leg raising: to raise the legs of the patients by adjusting the angle of the patient's bed during one minute.
  Tidal volume challenge: an increas by 2ml/Kg of the tidal volume during one minute
  Other Names: tidal volume challenge
  Groups: preload responders

SUMMARY:
Background: Predicting preload responsiveness by using dynamic indicators before administering fluids to critically ill patients is nowadays routinely performed at the bedside. Unlike other dynamic indicators of preload responsiveness that require cardiac output monitoring, pulse pressure variation (PPV) can be simply obtained via an arterial catheter . However, PPV is not reliable in mechanically ventilated patients with spontaneous breathing activity. We hypothesized that an increase in PPV after a tidal volume (TV) challenge (TVC) or a decrease in PPV during passive leg raising (PLR) will predict preload responsiveness in such cases.

Objective: to examine if the change in PPV during PLR and after a TVC can predict preload responsiveness in patients with mechanical ventilation and persistent spontaneous breathing

DETAILED DESCRIPTION:
Prospective non interventional study conducted in two intensive care units. Patients under mechanical ventilation with spontaneous cycles, for whom the physician in charge decided to test preload responsiveness were included. We collected demographic and clinical information, the use of mechanical ventilation and its parameters, the use of vasopressors and their dosage and blood lactate.

Firstly, transthoracic echocardiography (TTE) was performed to measure the velocity time integral (VTI) of the left ventricular outflow tract .

A PLR maneuvre is performed with TTE probe in place and a new assessement of VTI is measured, in addition to the PPV and other hemodynamic parmeters (Diastolic, mean and systolic arterial pressure, heart rate, CVP). Delta VTI is the difference between VTI during PLR and VTI at baseline divided by VTI at baseline.

Patients were considered as preload responsive when delta VTI was ≥10%. Secondly, a TVC was performed by increasing the TV by 2mL/kg predicted body weight from its baseline value . PPV was recorded before and after the TVC in addition to the other hemodynamic parmeters listed above. Further more, respiratory parameters are collected: ventilator setting, plateau pressure, upper airway pressure, before and during the TVC.

ELIGIBILITY:
Inclusion Criteria:

* adult critically ill patients if the clinicians in charge decided to test preload responsiveness because of mean arterial pressure (MAP) < 65 mmHg (measured by an arterial catheter) or other symptoms of acute circulatory failure (e.g. oliguria, skin mottling, tachycardia, hyperlactatemia)

Exclusion Criteria:

* Arrythmia
* no spontaneous breathing
* difficult condition for tansthoracic echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under mechanical ventilation with spontaneous cycles, for whom the physician in charge decided to test preload responsiveness were included with because of mean arterial pressure (MAP) < 65 mmHg (measured by an arterial catheter) or other symptoms of acute circulatory failure (e.g. oliguria, skin mottling, tachycardia, hyperlactatemia)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
predictive capacity of the changes of PPV during tidal volume challenge | duration of the tests: 15 minutes
  A roc curve analysis will be performed in order to determine the specificity and the sensitivity of this test to predict preload responsiveness

SECONDARY OUTCOMES:
predictive capacity of changes of PPV during ppassive leg raising test | duration of the tests: 15 minutes
  A roc curve analysis will be erformed in order to determine the specificity and the sensitivity of this test to predict preload responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Hamzaoui Olfa, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi R, Moretto F, Prat D, Jacobs F, Teboul JL, Hamzaoui O. Dynamic changes of pulse pressure but not of pulse pressure variation during passive leg raising predict preload responsiveness in critically ill patients with spontaneous breathing activity. J Crit Care. 2022 Dec;72:154141. doi: 10.1016/j.jcrc.2022.154141. Epub 2022 Sep 15. PMID 36116288
- [Derived] Hamzaoui O, Shi R, Carelli S, Sztrymf B, Prat D, Jacobs F, Monnet X, Gouezel C, Teboul JL. Changes in pulse pressure variation to assess preload responsiveness in mechanically ventilated patients with spontaneous breathing activity: an observational study. Br J Anaesth. 2021 Oct;127(4):532-538. doi: 10.1016/j.bja.2021.05.034. Epub 2021 Jul 8. PMID 34246460